CLINICAL TRIAL: NCT05270954
Title: Randomized, Double-blind, Multicenter Parallel-group Clinical Study of Safety, Tolerability and Immunogenicity of the Betuvax-CoV-2 Recombinant COVID-19 Vaccine, Suspension for Intramuscular Administration in Healthy Adult Volunteers
Brief Title: Safety, Tolerability and Immunogenicity of Recombinant COVID-19 Vaccine Betuvax-CoV-2
Acronym: Betuvax-CoV2
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Artgen Biotech (Other)
Collaborators: Betuvax LLC (Unknown); CEG BIO LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Betuvax-CoV-2.2021.CT1-2.RUS
Record Dates: First submitted 2022-03-02; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; coronavirus; recombinant vaccine; virus-like vaccine; betulin
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Phase 1 is Open Label; The Phase 2 is double-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (Phase 1) (Active Comparator): All volunteers randomized to Group 1 will be administered the Betuvax-CoV-2 drug according to the following scheme: 20 μg + 5 μg, twice, within a 28-day period.
  Interventions: Biological: Betuvax-CoV-2
- Group 2 (Phase 1) (Active Comparator): All volunteers randomized to Group 2 will be administered the Betuvax-CoV-2 drug according to the following scheme: 20 μg + 20 μg, twice, within a 28-day period.
  Interventions: Biological: Betuvax-CoV-2
- Group 3 (Phase 2) (Active Comparator): All volunteers randomized to Group 3 will be administered the Betuvax-CoV-2 drug according to the following scheme: 20 μg + 5 μg, twice, within a 28-day period.
  Interventions: Biological: Betuvax-CoV-2
- Group 4 (Phase 2) (Active Comparator): All volunteers randomized to Group 4 will be administered the Betuvax-CoV-2 drug according to the following scheme: 20 μg + 20 μg, twice, within a 28-day period.
  Interventions: Biological: Betuvax-CoV-2
- Group 5 (Phase 2) (Placebo Comparator): Volunteers randomized to Group 5 will be administered a placebo reference drug (0.9% aqueous sodium chloride solution), twice, within a 28-day period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Betuvax-CoV-2 — Vaccine: Betuvax-CoV-2 intramuscular injection solution (0.5 ml)
  Arms: Group 1 (Phase 1); Group 2 (Phase 1); Group 3 (Phase 2); Group 4 (Phase 2)
Drug: Placebo — Placebo: a 0.9% NaCl intramuscular injection solution (0.5 ml)
  Other Names: 0.9% NaCl
  Arms: Group 5 (Phase 2)

SUMMARY:
Randomized, double-blind, multicenter parallel-group clinical study of safety, tolerability and immunogenicity of the Betuvax-CoV-2 vaccine. The aim of this study is to investigate the safety, tolerability and immunogenicity of the Betuvax-CoV-2 Recombinant vaccine for the prevention of coronavirus infection caused by the SARS-CoV-2 virus, suspension for intramuscular administration, 10 μg/ml and 40 μg/ml (Ltd. Institute of New Medical Technologies, Russia) in healthy adult volunteers, aged 18 to 60 (inclusive).

DETAILED DESCRIPTION:
Participation of the volunteers in the study includes Visit 0 (screening), Visits 1-4 and Visits 10-13 (on an inpatient basis), Visits 5-9 and Visits 14-20 (on an outpatient basis). During Visits 2 and 11, volunteers receive either a study drug (one of two dosages) or a placebo.

The study includes 116 healthy male and female volunteers aged 18 to 60 (inclusive) years who meet the inclusion criteria.

All volunteers are enrolled in two stages of the study and at each stage they are randomized into two or three groups, respectively.

Taking into account the estimated number of volunteers found by the screening results as not meeting the inclusion criteria (54 people), 170 volunteers are screened in the First and Second stage.

The vaccination course includes two intramuscular injections within a 28-day period.

The first stage of the study:

* Group 1 (10 people) will be intramuscularly administered the study drug Betuvax-CoV-2 according to the following scheme: the first injection of 20 μg (0.5 ml of suspension for intramuscular administration of 40 μg/ml), the second injection of 5 μg (0.5 ml of suspension for intramuscular injection of 10 μg/ml) in 28 days.
* Group 2 (10 people) will be intramuscularly administered the study drug Betuvax-CoV-2 according to the following scheme: the first and second injection of 20 μg (0.5 ml of solution for intramuscular injection of 40 μg/ml) within a 28-day period.

The second stage of the study:

* Group 3 (32 people) will be intramuscularly administered the study drug Betuvax-CoV-2 according to the following scheme: the first injection of 20 μg (0.5 ml of the suspension for intramuscular administration of 40 μg/ml), the second injection of 5 μg (0.5 ml of the suspension for intramuscular injection of 10 μg/ml) in 28 days.
* Group 4 (32 people) will be intramuscularly administered the study drug Betuvax-CoV-2 according to the following scheme: the first and second injection of 20 μg (0.5 ml of solution for intramuscular injection of 40 μg/ml) within a 28-day period.
* Group 5 (32 people) will receive a placebo according to the following scheme: the first and second injections (0.5 ml of sodium chloride 0.9% solution, intramuscularly) within a 28-day period.

Study participants will be closely monitored for their intended outcomes. Key safety outcomes will be centrally reviewed by the Independent Data Monitoring Committee (ICMD). Investigators will be required to report anticipated safety outcomes in a timely manner (within 24 hours if possible) and to record these outcomes in the CRF in a timely manner (within 24 hours if possible).

ELIGIBILITY:
Inclusion criteria:

1. 18 to 60 years of age.
2. Verified healthy condition according to the data of standard clinical, laboratory and instrumental examination methods.
3. For women being in an active reproductive period: Consent to adhere to appropriate methods of contraception during the entire period of the participation in the study and for 1 month after the completion of the participation in the study (appropriate methods of contraception include abstinence from sexual intercourse or any two of the following methods: an intrauterine device (intrauterine device without release and with a release of a local hormonal drug), diaphragm, spermicides, cervical caps, oral contraceptives, contraceptive sponge and/or condom); for men: Consent to adhere to appropriate dual barrier methods of contraception during the entire period of the participation in the study and 1 month after completion of the participation in the study.
4. Body mass index (BMI): 18.5≤ BMI≤30 kg/m2.
5. Negative breath alcohol test.
6. Negative laboratory blood tests for HIV, syphilis and hepatitis B and C.
7. Ability and willingness to attend all scheduled visits and undergo all procedures and examinations planned by the Protocol.
8. Signed and dated Informed Consent to participate in the study.

Exclusion criteria:

1. Contact with COVID-19 patients during 14 days before the start of the study.
2. PCR SARS-CoV-2 positive test.
3. Titer of the total specific anti-SARS-CoV-2 antibodies (ELISA) more than 1:10.
4. Drug allergies, hereditary angioedema.
5. Hypersensitivity to any component of the vaccine or any excipients of Betuvax-CoV-2 or allergy to the components of the vaccine.
6. Intolerance to any of the components or any excipients of the vaccine Betuvax-CoV-2.
7. Allergic reaction to previous immunizations.
8. Serious post-vaccination reactions/complications associated with previous immunizations.
9. For women of childbearing potential - lactation period, pregnancy or suspicion of it, early postpartum period.
10. Women in the premenopausal period (last menstrual period <1 year prior to signing informed consent) who are not surgically sterile and women who have childbearing potential but do not use or plan to use appropriate methods of contraception throughout the study and do not agree to perform a urine pregnancy test while participating in a study.
11. Men who serve in the military by conscription.
12. Individuals in custody in pre-trial detention centers and those serving sentences in places of deprivation of liberty.
13. Children under 18 years of age.
14. Chronic diseases (including oncological and autoimmune), diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as the gastrointestinal tract, liver, kidneys, blood, central nervous system; surgical interventions on the gastrointestinal tract (with the exception of appendectomy).
15. Active tuberculosis at the time of screening (based on history and physical examination).
16. Mental illness, current or in history.
17. Decompensated neuropsychiatric diseases, including schizophrenia, multiple sclerosis, Parkinson's disease, dementia, endogenous depression, etc., which complicate the participation of a volunteer in the study.
18. Acute infectious from less than 3 months before the start of the study.
19. Acute infectious or non-infectious diseases, exacerbation of chronic diseases from less than 4 weeks before the start of the study.
20. Symptoms of any diseases at the time of enrollment or if less than 4 weeks have passed since recovery.
21. Hepatic or renal failure, currently or in history.
22. Current or history of oncological diseases.
23. Major surgery, major trauma less than 6 months prior to study initiation.
24. History of splenectomy.
25. Other comorbidities that, in the opinion of the investigator, may interfere with the evaluation of the objectives of the study.
26. Blood pressure: systolic blood pressure less than 100 mmHg or above 130 mmHg and diastolic blood pressure over 90 mmHg or less than 70 mmHg.
27. Heart rate less than 60 beats/min or more than 90 beats/min.
28. Deviations from the normal values according to standard clinical, laboratory (general and biochemical blood tests, urinalysis) and instrumental methods (including ECG) examination.
29. Long-term use (more than 14 days) of immunosuppressants, systemic glucocorticosteroids or immunomodulatory drugs during the 6 months before the start of the study.
30. Any vaccination within one month prior to the start of the clinical trial.
31. Taking medications containing immunoglobulin or blood products during the last 3 months before the start of the study.
32. Donation of blood (450 ml of blood or plasma and more) less than 2 months before the start of the study.
33. Participation in another clinical study less than 3 months before the start of the study.
34. Consumption of more than 10 units of alcohol (1 unit of alcohol is equivalent to 1/2 liter of beer, 200 ml of wine or 50 ml of spirits) per week or history of alcoholism, drug addiction, drug abuse.
35. Smoking more than 10 cigarettes a day.
36. Special diet (for example, vegetarian, vegan, with limited salt intake) or a special lifestyle (work at night, extreme physical activity).
37. Positive urine test result for psychotropic and narcotic substances, psychoactive drugs (barbiturates, benzodiazepines, methadone, phencyclidine).
38. Unwillingness or inability to follow the recommendations and procedures prescribed by this protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-04-25 (Estimated); Study Completion 2022-07-24 (Estimated)

PRIMARY OUTCOMES:
Total specific anti-SARS-CoV-2 antibodies | 21 days after the second administration of the study drug/placebo
  The proportion of the volunteers with an increased level of the total specific anti-SARS-CoV-2 antibodies by 4 times or more (ELISA test)
Total specific anti-SARS-CoV-2 antibodies | 90±5 days after the first administration of the study drug/placebo
  The proportion of the volunteers with an increased level of the total specific anti-SARS-CoV-2 antibodies by 4 times or more (ELISA test)
Neutralizing anti-SARS-CoV-2 antibodies | 21 days after the second administration of the study drug/placebo
  The proportion of the volunteers tested positive for the presence of neutralizing anti-SARS-CoV-2 antibodies (SARS-CoV-2 Surrogate Virus Neutralization Test)
Neutralizing anti-SARS-CoV-2 antibodies | 90±5 days after the first administration of the study drug/placebo
  The proportion of the volunteers tested positive for the presence of neutralizing anti-SARS-CoV-2 antibodies (SARS-CoV-2 Surrogate Virus Neutralization Test)
Adverse events | Within 50 days of the first dose of the study drug/placebo
  The proportion of the volunteers with any adverse events
Severe adverse events | Within 50 days of the first dose of the study drug/placebo
  The proportion of the volunteers with severe adverse events

SECONDARY OUTCOMES:
Total specific anti-SARS-CoV-2 antibodies | 180±5 days after the first administration of the study drug/placebo
  The proportion of the volunteers with an increased level of the total specific anti-SARS-CoV-2 antibodies by 4 times or more (ELISA test)
IgG-specific anti-SARS-CoV-2 antibodies | 21 days after the second administration of the study drug/placebo
  The proportion of the volunteers with an increased level of the IgG-specific anti-SARS-CoV-2 antibodies by 4 times or more (ELISA test)
IgG-specific anti-SARS-CoV-2 antibodies | 90±5 days after the first dose of the study drug/placebo
  The proportion of the volunteers with an increased level of the IgG-specific anti-SARS-CoV-2 antibodies by 4 times or more (ELISA test)
IgG-specific anti-SARS-CoV-2 antibodies | 180±5 days after the first dose of the study drug/placebo
  The proportion of the volunteers with an increased level of the IgG-specific anti-SARS-CoV-2 antibodies by 4 times or more (ELISA test)
IgM-specific anti-SARS-CoV-2 antibodies | 21 days after the second administration of the study drug/placebo
  The proportion of the volunteers with an increased level of the IgM-specific anti-SARS-CoV-2 antibodies by 4 times or more (ELISA test)
IgM-specific anti-SARS-CoV-2 antibodies | 90±5 days after the first dose of the study drug/placebo
  The proportion of the volunteers with an increased level of the IgM-specific anti-SARS-CoV-2 antibodies by 4 times or more (ELISA test)
IgM-specific anti-SARS-CoV-2 antibodies | 180±5 days after the first dose of the study drug/placebo
  The proportion of the volunteers with an increased level of the IgM-specific anti-SARS-CoV-2 antibodies by 4 times or more (ELISA test)
Neutralizing anti-SARS-CoV-2 antibodies | 180±5 days after the first administration of the study drug/placebo
  The proportion of the volunteers tested positive for the presence of neutralizing anti-SARS-CoV-2 antibodies (SARS-CoV-2 Surrogate Virus Neutralization Test)
Geometric mean titers of the total anti-SARS-CoV-2 antibodies | 21 days after the second administration of the study drug/placebo
  The proportion of the volunteers with geometric mean titers of the total anti-SARS-CoV-2 antibodies (ELISA test)
Geometric mean titers of the total anti-SARS-CoV-2 antibodies | 90±5 days after the first administration of the study drug/placebo
  The proportion of the volunteers with geometric mean titers of the total anti-SARS-CoV-2 antibodies (ELISA test)
Geometric mean titers of the total anti-SARS-CoV-2 antibodies | 180±5 days after the first administration of the study drug/placebo
  The proportion of the volunteers with geometric mean titers of the total anti-SARS-CoV-2 antibodies (ELISA test)
Geometric mean titers of the IgG-specific anti-SARS-CoV-2 antibodies | 21 days after the second administration of the study drug/placebo
  The proportion of the volunteers with geometric mean titers of the IgG-specific anti-SARS-CoV-2 antibodies (ELISA test)
Geometric mean titers of the IgG-specific anti-SARS-CoV-2 antibodies | 90±5 days after the first administration of the study drug/placebo
  The proportion of the volunteers with geometric mean titers of the IgG-specific anti-SARS-CoV-2 antibodies (ELISA test)
Geometric mean titers of the IgG-specific anti-SARS-CoV-2 antibodies | 180±5 days after the first administration of the study drug/placebo
  The proportion of the volunteers with geometric mean titers of the IgG-specific anti-SARS-CoV-2 antibodies (ELISA test)
Geometric mean titers of the IgM-specific anti-SARS-CoV-2 antibodies | 21 days after the second administration of the study drug/placebo
  The proportion of the volunteers with geometric mean titers of the IgM-specific anti-SARS-CoV-2 antibodies (ELISA test)
Geometric mean titers of the IgM-specific anti-SARS-CoV-2 antibodies | 90±5 days after the first administration of the study drug/placebo
  The proportion of the volunteers with geometric mean titers of the IgM-specific anti-SARS-CoV-2 antibodies (ELISA test)
Geometric mean titers of the IgM-specific anti-SARS-CoV-2 antibodies | 180±5 days after the first administration of the study drug/placebo
  The proportion of the volunteers with geometric mean titers of the IgM-specific anti-SARS-CoV-2 antibodies (ELISA test)
Specific anti-SARS-CoV-2 cellular immune response (Phase 1) | 21 days after the second dose of the study drug (only in Phase 1)
  The proportion of the volunteers with a specific anti-SARS-CoV-2 cellular immune response (flow cytometry)
Specific anti-SARS-CoV-2 cellular immune response (Phase 1) | 90±5 days after the first dose of the study drug (only in Phase 1)
  The proportion of the volunteers with a specific anti-SARS-CoV-2 cellular immune response (flow cytometry)
Specific anti-SARS-CoV-2 cellular immune response | 21 days after the second dose of the study drug/placebo
  The proportion of the volunteers with a specific anti-SARS-CoV-2 cellular immune response (ELISPOT)
Specific anti-SARS-CoV-2 cellular immune response | 90±5 days after the first dose of the study drug/placebo
  The proportion of the volunteers with a specific anti-SARS-CoV-2 cellular immune response (ELISPOT)
Specific anti-SARS-CoV-2 cellular immune response | 180±5 days after the first dose of the study drug/placebo
  The proportion of the volunteers with a specific anti-SARS-CoV-2 cellular immune response (ELISPOT)
COVID-19 symptoms | From the 7th day after the second administration of the study drug/placebo till the 90±5 day after the first dose of study drug/placebo
  The proportion of the volunteers with at least one COVID-19 symptom (fever, chills, dyspnoea, difficulty breathing, cough, sore throat, fatigue, muscle pain, loss or decrease in taste and/or odor, nasal congestion, runny nose, headache, nausea, vomiting, diarrhea) and a PCR-confirmed SARS-CoV-2 infection
COVID-19 symptoms | From the 7th day after the second administration of the study drug/placebo till the 180±5 day after the first dose of study drug/placebo
  The proportion of the volunteers with at least one COVID-19 symptom (fever, chills, dyspnoea, difficulty breathing, cough, sore throat, fatigue, muscle pain, loss or decrease in taste and/or odor, nasal congestion, runny nose, headache, nausea, vomiting, diarrhea) and a PCR-confirmed SARS-CoV-2 infection
Moderate, severe or extremely severe course of COVID-19, or lethal outcome | From the 7th day after the second administration of the study drug/placebo till the 90±5 day after the first dose of the study drug/placebo
  The proportion of the volunteers with COVID-19 of moderate, severe or extremely severe course, or with a lethal outcome, and a PCR-confirmed SARS-CoV-2 infection
Moderate, severe or extremely severe course of COVID-19, or lethal outcome | From the 7th day after the second administration of the study drug/placebo till the 180±5 day after the first dose of the study drug/placebo
  The proportion of the volunteers with COVID-19 of moderate, severe or extremely severe course, or with a lethal outcome, and a PCR-confirmed SARS-CoV-2 infection
Severe or extremely severe course of COVID-19, or lethal outcome | From the 7th day after the second administration of the study drug/placebo till the 90±5 day after the first dose of the study drug/placebo
  The proportion of the volunteers with COVID-19 of severe or extremely severe course, or with a lethal outcome, and a PCR-confirmed SARS-CoV-2 infection
Severe or extremely severe course of COVID-19, or lethal outcome | From the 7th day after the second administration of the study drug/placebo till the 180±5 day after the first dose of the study drug/placebo
  The proportion of the volunteers with COVID-19 of severe or extremely severe course, or with a lethal outcome, and a PCR-confirmed SARS-CoV-2 infection
Lethal outcome | From the 7th day after the second administration of the study drug/placebo till the 90±5 day after the first dose of the study drug/placebo
  The proportion of the volunteers with lethal outcome, and a PCR-confirmed SARS-CoV-2 infection
Lethal outcome | From the 7th day after the second administration of the study drug/placebo till the 180±5 day after the first dose of the study drug/placebo
  The proportion of the volunteers with lethal outcome, and a PCR-confirmed SARS-CoV-2 infection
Allergic reactions | Within 2 hours of the first study drug/placebo administration
  The proportion of the volunteers with immediate side effects (allergic reactions)
Allergic reactions | Within 2 hours of the second study drug/placebo administration
  The proportion of the volunteers with immediate side effects (allergic reactions)
Local post-vaccination reactions | Within 7 days after the first administration of the study drug/placebo
  The proportion of the volunteers with local post-vaccination reactions
Local post-vaccination reactions | Within 7 days after the second administration of the study drug/placebo
  The proportion of the volunteers with local post-vaccination reactions
Severe local post-vaccination reactions | Within 7 days of the first study drug/placebo administration
  The proportion of the volunteers with >grade 3 of local post-vaccination reactions
Severe local post-vaccination reactions | Within 7 days of the second study drug/placebo administration
  The proportion of the volunteers with >grade 3 of local post-vaccination reactions
Systemic post-vaccination reactions | Within 7 days after the first administration of the study drug/placebo
  The proportion of the volunteers with systemic post-vaccination reactions
Systemic post-vaccination reactions | Within 7 days after the second administration of the study drug/placebo
  The proportion of the volunteers with systemic post-vaccination reactions
Severe systemic post-vaccination reactions | Within 7 days after the first administration of the study drug/placebo
  The proportion of the volunteers with >grade 3 of severe systemic post-vaccination reactions
Severe systemic post-vaccination reactions | Within 7 days after the second administration of the study drug/placebo
  The proportion of the volunteers with >grade 3 of severe systemic post-vaccination reactions
Any adverse events | Within 90±5 days after the first dose of the study drug/placebo
  The proportion of the volunteers with any adverse events
Any adverse events | Within 180±5 days after the first dose of the study drug/placebo
  The proportion of the volunteers with any adverse events
Adverse events of special interest | Within 50 days after the first dose of the study drug/placebo
  The proportion of the volunteers with adverse events of special interest, adverse reactions that require medical attention, with newly developed chronic diseases
Adverse events of special interest | Within 90±5 days after the first dose of the study drug/placebo
  The proportion of the volunteers with adverse events of special interest, adverse reactions that require medical attention, with newly developed chronic diseases
Adverse events of special interest | Within 180±5 days after the first dose of the study drug/placebo
  The proportion of the volunteers with adverse events of special interest, adverse reactions that require medical attention, with newly developed chronic diseases
Severe adverse events | Within 90±5 days after the first dose of the study drug/placebo
  The proportion of the volunteers with severe adverse events
Severe adverse events | Within 180±5 days after the first dose of the study drug/placebo
  The proportion of the volunteers with severe adverse events
Prematurely terminated participation | Within 50 days after the administration of the first dose of the study drug/placebo
  The proportion of the volunteers who prematurely terminated their participation in the study due to the development of adverse events or severe adverse events associated with the use of the study drug
Prematurely terminated participation | Within 90±5 days after the administration of the first dose of the study drug/placebo
  The proportion of the volunteers who prematurely terminated their participation in the study due to the development of adverse events or severe adverse events associated with the use of the study drug
Prematurely terminated participation | Within 180±5 days after the administration of the first dose of the study drug/placebo
  The proportion of the volunteers who prematurely terminated their participation in the study due to the development of adverse events or severe adverse events associated with the use of the study drug

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Center of professional medicine, Perm
  - "Eco-Safety" R&D center, Saint Petersburg
  - Department of Vaccinology, Smorodintsev Research Institute of Influenza of the Ministry of Health of the Russian Federation, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kudriavtsev AV, Vakhrusheva AV, Kryuchkov NA, Frolova ME, Blagodatskikh KA, Ivanishin TV, Djonovic M, Romanovskaya-Romanko EA, Kovalenko AN, Lioznov DA, Zubkova TG, Teplykh SV, Oseshnyuk RA, Stukova MA, Isaev AA, Krasilnikov IV. Safety and Immunogenicity of Betuvax-CoV-2, an RBD-Fc-Based SARS-CoV-2 Recombinant Vaccine: Preliminary Results of the First-in-Human, Randomized, Double-Blind, Placebo-Controlled Phase I/II Clinical Trial. Vaccines (Basel). 2023 Feb 1;11(2):326. doi: 10.3390/vaccines11020326. PMID 36851204